CLINICAL TRIAL: NCT07395245
Title: Mental Health Literacy and Help-Seeking Behavior Among Adolescents in Assiut City: An Interventional Study
Brief Title: Mental Health Literacy and Help-Seeking Behavior Among Adolescents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mireille Maged Emile Hanna, Assistant Lecturer at the Public Health Department, Faculty of Medicine, Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Mental Health in Adolescents
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Mental Health; Mental Health Literacy; Stigma of Mental Illness; Help-Seeking Behavior; Adolescent Mental Health
Keywords: Mental Health Literacy; Help-Seeking Behavior; Adolescent Mental Health; Stigma
MeSH Terms: conditions — Psychological Well-Being; Help-Seeking Behavior; Social Stigma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental Health Literacy Educational Program (Experimental): Participants receive a brief school-based educational intervention consisting of three structured classroom sessions delivered over 3 consecutive weeks. Session 1 covers mental health literacy (basic concepts, common adolescent mental health problems, signs/symptoms, myths vs facts). Session 2 addresses stigma reduction (public stigma, self-stigma, respectful language). Session 3 focuses on help-seeking behavior (informal vs formal help sources, barriers, local resources in Assiut, role-play activities). Each session includes 30-40 minutes of teaching plus 10 minutes of discussion/activities. Pre-test and post-test assessments (MHLS, PMHSS, GHSQ, ATSPPH, SDQ) are administered before the intervention and 1 month after completion.
  Interventions: Behavioral: School-Based Mental Health Literacy Educational Program
- No Intervention Control (No Intervention): Participants receive no educational intervention during the study period. They continue with their regular school activities without any mental health literacy sessions. Pre-test and post-test assessments using the same validated questionnaires (Mental Health Literacy Scale, Peer Mental Health Stigmatization Scale, General Help-Seeking Questionnaire, Attitudes Toward Seeking Professional Psychological Help scale, and Strengths and Difficulties Questionnaire) are administered at the same time points as the intervention group: before the intervention period begins and 1 month after the intervention group completes the three sessions.

INTERVENTIONS:
Behavioral: School-Based Mental Health Literacy Educational Program — A school-based educational program delivered over 3 consecutive weeks, consisting of three 40-50 minute structured classroom sessions. Session 1 (Mental Health Literacy) covers basic concepts of mental health and mental illness, common adolescent mental health problems including stress, anxiety, and depression, key signs and symptoms, and myths versus facts about mental health. Session 2 (Stigma Reduction) addresses what stigma is, how negative labels and stereotypes affect people with mental health problems, differences between public stigma and self-stigma, and promotes respectful language through interactive activities. Session 3 (Help-Seeking Behavior) focuses on recognizing when problems need help, differences between informal and formal help sources, common barriers to seeking help, and provides information about local mental health resources in Assiut including role-play activities on how to approach trusted adults.
  Arms: Mental Health Literacy Educational Program

SUMMARY:
This study examines mental health awareness and help-seeking behaviors among adolescents aged 13-18 years in Assiut City, Egypt. Mental health problems are common among young people, but many adolescents do not seek professional help when they need it. This is often due to low mental health literacy (not understanding mental health problems or knowing where to get help), stigma (negative attitudes toward mental illness), and fears about confidentiality or being judged.

The study has two parts:

Part 1 - Assessment Phase: Researchers will survey approximately 270 students from preparatory and secondary schools in Assiut to understand their current levels of mental health literacy, stigma, and willingness to seek help for mental health problems. Students will complete validated questionnaires that measure their knowledge about mental health, their attitudes toward peers with mental health problems, and their intentions to seek help from various sources.

Part 2 - Intervention Phase: In a randomized controlled trial involving 150 students (75 in an intervention group and 75 in a control group), researchers will test whether a brief educational program can improve mental health literacy, reduce stigma, and increase help-seeking intentions. The intervention consists of three weekly classroom sessions covering: (1) mental health literacy - basic concepts, common problems in adolescents like stress and anxiety, recognizing symptoms; (2) stigma reduction - understanding how negative labels hurt people, recognizing public and self-stigma, using respectful language; and (3) help-seeking behavior - knowing when to seek help, understanding formal and informal help sources, overcoming barriers, and learning about local resources in Assiut.

Students in both groups will complete questionnaires before the intervention and one month after completion. The control group will not receive the educational sessions during the study period. Researchers will compare changes in mental health knowledge, stigma levels, and help-seeking attitudes between the two groups to determine whether the program is effective.

The study aims to address a critical gap in mental health services for adolescents in Upper Egypt by improving young people's understanding of mental health and encouraging them to seek appropriate help when needed.

DETAILED DESCRIPTION:
Background and Rationale:

Mental health problems among adolescents represent a significant public health burden worldwide and in Egypt. Studies among Egyptian secondary school and university students show high prevalence of depression (32.5%), anxiety (45.2%), and psychological distress (65-70%). Despite this burden, most adolescents do not seek professional help due to low mental health literacy, stigma, and lack of awareness of available services. Existing Egyptian research focuses primarily on urban university students, leaving a critical evidence gap for younger school-aged adolescents, particularly in underserved regions like Upper Egypt.

Study Design:

This is a two-phase study combining cross-sectional assessment and a randomized controlled trial.

Phase 1 - Cross-Sectional Assessment (n=270):

Four preparatory/secondary schools in Assiut city will be randomly selected using cluster sampling stratified by educational stage and school gender composition. All eligible students aged 13-18 years will be invited to complete validated Arabic questionnaires assessing mental health literacy (MHLS - 35 items covering six domains), peer stigmatization (PMHSS - 16 items), help-seeking intentions (GHSQ), attitudes toward professional help (ATSPPH - 10 items), and mental health difficulties (SDQ - 25 items). Sociodemographic data will also be collected. This phase establishes baseline prevalence and identifies factors associated with mental health literacy, stigma, and help-seeking patterns.

Phase 2 - Randomized Controlled Trial (n=150):

Two secondary schools (one male, one female) will be selected. Within each school, 75 students will be randomly assigned to the intervention group and 75 to the control group, matched for age and sex. The intervention consists of three weekly structured classroom sessions (40-50 minutes each) delivered by trained researchers:

Session 1 (Mental Health Literacy): Basic concepts of mental health and mental illness; common adolescent mental health problems including stress, anxiety, and depression; key signs and symptoms; myths versus facts about mental health; understanding that mental health problems are real, treatable conditions.

Session 2 (Stigma Reduction): Definition and impact of stigma; how negative labels and stereotypes harm people with mental health problems; distinction between public stigma (others' attitudes) and self-stigma (internalized shame); recognition of stigma in adolescent contexts (mocking, exclusion, gossip); activities promoting respectful language and empathy.

Session 3 (Help-Seeking Behavior): Recognizing when problems require professional help; differences between informal sources (family, friends, religious leaders) and formal/professional sources (school counselors, physicians, psychiatrists, youth health centers); common barriers to help-seeking including shame, fear, and confidentiality concerns; information about realistic, accessible mental health resources in Assiut; role-play exercises on approaching trusted adults and guiding peers to help.

All sessions use interactive teaching methods with clear examples, group discussions, and brief activities. The control group continues regular school activities without receiving intervention sessions during the study period. Both groups complete identical questionnaires at baseline and one month post-intervention.

Assessment Tools:

All instruments are validated Arabic versions: Mental Health Literacy Scale (MHLS), Peer Mental Health Stigmatization Scale (PMHSS), General Help-Seeking Questionnaire (GHSQ), Attitudes Toward Seeking Professional Psychological Help scale (ATSPPH), and Strengths and Difficulties Questionnaire (SDQ).

Expected Outcomes:

This study will provide the first comprehensive data on mental health literacy, stigma, and help-seeking among school-aged adolescents in Assiut and Upper Egypt. It will test whether a brief, feasible school-based intervention can improve knowledge, reduce stigma, and promote help-seeking behaviors, potentially informing scalable mental health promotion strategies for Egyptian schools.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 13-18 years.
* Enrolled in selected schools in Assiut city

Exclusion Criteria:

* Documented severe intellectual disability or learning difficulty that, in the judgement of school staff, would prevent understanding of the intervention content or valid questionnaire completion.
* Current acute medical or psychiatric emergency at the time of data collection as identified by school or health-center staff.
* Refusal of participation by the student, or absence of parental consent.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in Mental Health Literacy Scale (MHLS) Total Score | 1 month after completion of the intervention program
  Change in total score on the Mental Health Literacy Scale (MHLS), a validated 35-item Arabic questionnaire that measures knowledge and understanding of mental health disorders, including recognition of disorders, knowledge of professional help sources, knowledge of self-help strategies, attitudes promoting appropriate help-seeking, knowledge of prevention, and ability to find and use mental health information. Items are scored on Likert scales. Higher total scores indicate greater mental health literacy. Change is calculated as post-intervention score minus baseline score.

SECONDARY OUTCOMES:
Change in Peer Mental Health Stigmatization Scale (PMHSS) Score | 1 month after completion of the intervention program
  The Peer Mental Health Stigmatization Scale (PMHSS) is a validated 16-item Arabic questionnaire measuring adolescents' stigmatizing attitudes toward peers with mental health problems, including stereotypes, prejudice, and discrimination. Items are scored on a 5-point Likert scale, with higher scores indicating greater stigmatization. The outcome is the between-group difference in change scores comparing intervention versus control groups.